CLINICAL TRIAL: NCT00811915
Title: A Prospective, Comparative, Multicenter, Randomized Study to Compare the Safety and Efficacy of Sirolimus (Rapamune) to Tacrolimus (Advagraf) Associated to Mycophenolate Mofetil (CellCept) Between 12 and 36 Months After Kidney Transplantation
Brief Title: Study to Compare the Safety and Efficacy of Sirolimus (Rapamune) to Tacrolimus (Advagraf) Associated to Mycophenolate Mofetil (CellCept) Between 12 and 36 Months After Kidney Transplantation
Acronym: EPARGNE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2007/125/HP
Record Dates: First submitted 2008-12-18; First posted 2008-12-19 (Estimated); Last update posted 2014-06-19 (Estimated); Status verified 2014-06

CONDITIONS: Kidney Transplantation
Keywords: Sirolimus; Tacrolimus; Kidney transplantation; Kidney Transplant Recipients
MeSH Terms: interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sirolimus (Experimental): Group A : Sirolimus introduction and tacrolimus withdrawal
  * Tacrolimus : 33 % decrease of daily dose with complete withdrawal at day 14.
  * Sirolimus daily dose according to CYP3A5 genotype CYP3A5*1/*1 or *1/*3: 4 mg/d CYPY3A5*3/*3 : sirolimus 2 mg/j Adjusted to obtain a trough level between 6 and10 ng/ml
  Interventions: Drug: Sirolimus
- B (Active Comparator): Tacrolimus (Advagraf) dose to obtain a trough level between 4 and 10 ng/ml
  Interventions: Drug: Sirolimus

INTERVENTIONS:
Drug: Sirolimus — Sirolimus introduction and tacrolimus withdrawal
  Tacrolimus : 33 % decrease of daily dose with complete withdrawal at day 14. Sirolimus daily dose according to CYP3A5 genotype CYP3A5*1/*1 or *1/*3: 4 mg/d CYPY3A5*3/*3 : sirolimus 2 mg/j Adjusted to obtain a trough level between 6 and10 ng/ml

SUMMARY:
The use of tacrolimus in the long term as part of the immunosuppressive regimen after transplantation is associated to complications such as chronic nephrotoxicity, impaired glucose metabolism (diabetes mellitus) and an increase of the incidence of neoplasia. The conversion from a tacrolimus based therapy to a sirolimus based therapy associated with mycophenolate mofetil could improve the incidence of such complications. The aim of this study is to assess the risk/benefit ratio of this switch performed in stable renal transplant recipient between 12 months and 36 months after transplantation. The incidence of a composite endpoint (worsening of GFR evaluated by MDRD formula, incidence of cancer and diabetes) will be assessed 24 months after conversion.

DETAILED DESCRIPTION:
Two doses of Sirolimus will be evaluated accorded to the CYP 3A5 genotype. Patients carrying at least CYP 3A5 *1 allele will receive 4 mg per day whereas the others (CYP 3A5 *3/*3) will receive 2 mg.

ELIGIBILITY:
Inclusion Criteria:

* Recipient age ≥18 and ≤ 75 ans.
* Patients having received a first or second renal transplant from a cadaveric or living related donor between 12 and 24 months prior the inclusion.
* Peak panel reactive antibody (PRA) < 30 %
* Patients with a stable renal function during the 3 months prior to inclusion (variation of serum creatinine lower than 20 %)
* Creatinine clearance ≥ 40 ml/mn/1.73 m26.
* Patients receiving as a stable immunosuppressive treatment associating: Mycophenolate mofetil (MPA AUC > 30 mg.h/L) and Tacrolimus with a trough level > 4 ng/ml, with or without corticoids

Exclusion Criteria:

* Multiorgan recipients
* Patients receiving cyclosporine
* Pregnancy
* Recipients of ABO incompatible graft
* Use of other immunosuppressive drugs.
* Historical peak reactive antibody ≥ 30 %
* Past medical history of humoral rejection, 2 episodes of acute cellular rejection
* Past medical history of sub-clinical rejection on routine allograft biopsy
* Calculated creatinine clearance < 40 ml/mn/1.73 m2
* 24h proteinuria > 1 g/24H
* Patients with severe diarrhea
* HTLV1 or HIV positivity
* Known hypersensitivity to tacrolimus, mycophenolate mofetil, or sirolimus.
* Total white blood cells < 2500/mm3 or hemoglobin < 9 g/dl

Ages: 18 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2009-01; Primary Completion 2013-12 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
The incidence of a composite endpoint (worsening of GFR estimated with MDRD formula, incidence of cancer and incidence of post-transplant diabetes mellitus) will be assessed 24 months after conversion. | 24 months

SECONDARY OUTCOMES:
*Renal function by calculated creatinine clearance* Incidence of biopsy proven acute rejection *Incidence of de novo diabetes mellitus *Incidence of hypertension *Incidence of skin cancer *Incidence of Chronic Rejection | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle ETIENNE, MD, Principal Investigator — University Hospital, Rouen
Locations (8):
- France (8):
  - UHAmiens, Amiens
  - UHAngers, Angers
  - UHCaen, Caen
  - UHLimoges, Limoges
  - UHNecker, Paris
  - UHRennes, Rennes
  - UHRouen, Rouen
  - UHTours, Tours